CLINICAL TRIAL: NCT01706705
Title: 3D Image-guided Intracavitary Brachytherapy Treatment Planning for Cervical Cancer Using a Novel Shielded Applicator
Brief Title: Magnetic Resonance Imaging (MRI) Brachytherapy Applicator Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2012-0546; NCI-2012-02120 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-10-11; First posted 2012-10-15 (Estimated); Results first posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-01

CONDITIONS: Cervical Cancer
Keywords: Cervical Cancer; Radiation therapy; XRT; External beam therapy; Brachytherapy; Intracavitary brachytherapy; ICBT; MRI compatible intracavitary applicators; Computed tomography; CT; Magnetic resonance imaging; MRI; MRI compatible applicators; 3D image guided treatment planning; 2D treatment planning
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brachytherapy Treatment Planning (Experimental): MRI-compatible intracavitary applicator inserted using ultrasound guidance to verify tandem placement in the uterus. Tandem and ovoids, tandem and cylinders, or tandem and ring chosen to accommodate patient's tumor and vaginal anatomy.
  Computed tomography (CT) scan and a magnetic resonance imaging (MRI) scan performed after the implant is placed in the operating room. The CT scan should take about 20 minutes and the MRI about 45 minutes.
  Interventions: Device: Intracavitary Applicator Placement; Other: Computed Tomography (CT); Other: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Device: Intracavitary Applicator Placement — MRI-compatible applicator inserted using ultrasound guidance to verify tandem placement in the uterus. Tandem and ovoids, tandem and cylinders, or tandem and ring chosen to accommodate patient's tumor and vaginal anatomy.
  Other Names: MDA Applicator
Other: Computed Tomography (CT) — CT scan performed after implant is placed in operating room. CT scan should take about 20 minutes.
  Other Names: CT
Other: Magnetic Resonance Imaging (MRI) — MRI scan performed after implant is placed in the operating room. MRI should take about 45 minutes.
  Other Names: MRI

SUMMARY:
The goal of this clinical research study is to learn if computed tomography (CT) and magnetic resonance imaging (MRI) images can better help to plan internal radiation treatment.

DETAILED DESCRIPTION:
Treatment planning for patients with cervical cancer treated at MD Anderson is usually performed based on x-ray films taken while the patient is under anesthesia in the operating room. In this study, you will have an MRI and CT scan performed after recovering from anesthesia in addition to the standard x-rays. In order to allow MRI images to be taken, special MRI compatible applicators will be used. The CT and MRI images will be reviewed by the doctor in charge of radiation treatment and will also be used for research purposes.

Study Procedures:

If you agree to take part in this study, an applicator made of a material that can be used during an MRI will be used.

You will have a CT scan and an MRI scan performed after the implant is placed in the operating room. The CT scan should take about 20 minutes and the MRI about 55 minutes. These scans will be performed after you wake up from general anesthesia. Pain medicine will be given if you feel any discomfort from the placement of the implant.

The additional scans will be used to confirm appropriate placement of the applicator and may result in small adjustments to your radiation treatment plan.

Length of Study:

Your active participation on this study will be complete once you have the CT and MRI scans.

Your medical record may be reviewed after the scans for the purposes of the study, but you will not be contacted in the future.

This is an investigational study. The applicator that best fits your personal anatomy will be used in this study. A selection of MRI compatible applicators are available. Many of the MRI applicators that will be used are FDA approved. However, in some cases you may have a novel device with a moveable shield placed. This applicator is not FDA approved or commercially available.

Up to 57 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1) Women with stage greater than or equal to IB2 cervical cancer treated with definitive chemoradiation or radiation therapy who require intracavitary brachytherapy.

Exclusion Criteria:

1. Patient or tumor anatomy that requires use of a non-MRI-compatible applicator.
2. Patients who require interstitial brachytherapy.
3. Patients whose treating physician feels that they require additional 3D imaging at the time of implant based on physical exam or initial findings.
4. Patients with implantable cardioverter-defibrillator, pacemaker or other implanted device, which precludes MRI acquisition.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2012-10-22 (Actual); Primary Completion 2018-04-22 (Actual); Study Completion 2018-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Klopp, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Brachytherapy Treatment Planning: Single Arm in which eligible patients were women with a diagnosis of 1B2cervical cancer with definitive chemoradiation or radiation therapy who required brachytherapy.
Period: Overall Study
Arm/Group | Experimental Brachytherapy Treatment Planning
Started | 57
Completed | 37
Not Completed | 20
Not completed — Death | 1
Not completed — Lack of Efficacy | 13
Not completed — Non-clinical | 6

BASELINE CHARACTERISTICS:
Arm/Group | Experimental Brachytherapy Treatment Planning
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 40 [25 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 34
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Improved Image Quality in the Shifted Position
Description: To determine the number of participants with improved image quality using the Novel Brachytherapy Applicator, using subjective and objective measures. In the subjective, for assessment of image quality for clinical use, the images obtained in the "shifted" position and in the "standard" position, were compared by a radiation oncologist without knowledge of which was the first and which was the second image. To provide and objective measure of the reduction in image artifact with the shields shifted, the bladder, rectum, and sigmoid were contoured, and average and standard deviation of Hounsfield units (HU) within these critical structures on the images were compared.
Time Frame: At the time of implant
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Brachytherapy Treatment Planning
Number analyzed (Participants) | 15
Participants
  Standard Position | 0
  Shifted Position | 15

2. Secondary Outcome: Number of Participants With High Quality Images With the Adaptive Applicator in the Shifted or Standard Position
Description: The number of participants with high quality images of the bladder, rectum and sigmoid with the adaptive applicator in the shifted position and standard position assessed by the Hounsfield unit values. The higher quality images are the images with higher density when the applicator is in either the shifted or standard position. The Hounsfield unit (HU) is a relative quantitative measurement of radio density used by radiologists in the interpretation of computed tomography (CT) images. The images obtained in the "shifted" position and in the "standard" position with the use of the adaptive applicator, were compared by a radiation oncologist without knowledge of which was the first and which was the second image.
Time Frame: At the time of implant
Population: The adaptive applicator fit into 15 of the evaluated patients so the analysis was limited to these 15 patients.
Measure: Count of Participants; unit: Participants
Groups:
- Single Arm-Study: Experimental Brachytherapy Treatment Planning
Arm/Group | Single Arm-Study
Number analyzed (Participants) | 15
Participants
  Adaptive Applicator in the Standard Position | 0
  Adaptive Applicator in the Shifted Position | 15

3. Other Pre Specified Outcome: 3D Image-guided Intracavitary Brachytherapy Treatment Planning in Cervical Cancer
Description: Analysis was conducted using JMP Pro statistical software for patients diagnosis of 1B2cervical cancer
Time Frame: 24 months from baseline
Population: No data collected
Arm/Group | Single Arm-Study
Number analyzed (Participants) | 0

4. Other Pre Specified Outcome: Magnetic Resonance Imaging (MRI) is Superior to Computed Tomography (CT) Imaging in Delineating a High Risk Target Volume. 3D Image-guided Intracavitary Brachytherapy Treatment Planning in Cervical Cancer".
Description: Utility of MRI imaging as compared to CT or MRI can improve dosimetric tumor coverage and normal tissue sparing.
Time Frame: 24 months from baseline ( 2-years)
Population: No data collected
Arm/Group | Single Arm-Study
Number analyzed (Participants) | 0

5. Other Pre Specified Outcome: Clinical and Tumor Characteristics of Patients in Whom CT or MRI Can Improve Dosimetric Tumor Coverage and Normal Tissue Sparing
Description: MRI-based brachytherapy planning for patients with tumors >5 cm and parametrial invasion on MRI at diagnosis and for those with a high BMI
Time Frame: 24 months from baseline ( 2-years)
Population: No data collected
Arm/Group | Single Arm-Study
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Feasibility of MRI-based Treatment Planning Utilizing the Shielded MD Anderson Adaptive Applicator.
Description: RI-adaptive applicators for treatment planning for every case/patient.
Time Frame: 24 months from baseline ( 2-years)
Population: No data collected
Arm/Group | Single Arm-Study
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Relative Resource Utilization for MRI and CT Based Treatment Planning as Compared to Standard Film Based Planning Techniques.
Description: Due to lack of a suitable comparison population during this timeframe- at our institution, these protocol-eligible cervical cancer patients were no longer undergoing brachytherapy treatment planning based solely off standard plain films alone.
Time Frame: Not able to complete
Population: Due to lack of a suitable comparison population during this timeframe- at our institution, these protocol-eligible cervical cancer patients were no longer undergoing brachytherapy treatment planning based solely off standard plain films alone.
Arm/Group | Single Arm-Study
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: At the time of implant
Groups:
- Experimental Brachytherapy Treatment Planning: Single Arm study in which eligible patients were women with a diagnosis of 1B2cervical cancer with definitive chemoradiation or radiation therapy who required brachytherapy.
Arm/Group | Experimental Brachytherapy Treatment Planning
All-Cause Mortality (participants affected / at risk) | 1/37
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-05-05): https://cdn.clinicaltrials.gov/large-docs/05/NCT01706705/Prot_SAP_000.pdf